CLINICAL TRIAL: NCT06986954
Title: Beacon Tip Sizing Catheter and Slip-Cath Beacon Tip Catheter Study
Status: Recruiting | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 24-01
Record Dates: First submitted 2025-05-08; First posted 2025-05-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Stenosis; Bleed Intracranial; Stroke; TIA; Vascular Malformation; Pseudoaneurysm
Keywords: Catheter; Beacon; Diagnostic imaging; Device sizing; Beacon tip slip cath
MeSH Terms: conditions — Constriction, Pathologic; Intracranial Hemorrhages; Stroke; Vascular Malformations; Aneurysm, False

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Beacon Tip Catheters: Beacon Tip Sizing Catheter and Slip-Catheter Beacon Tip Catheter & Shuttle Select Slip-Catheter (Visceral and Cerbral)
  Interventions: Device: Beacon Tip Catheters

INTERVENTIONS:
Device: Beacon Tip Catheters — Indicated for use in angiographic procedures by physicians trained and experienced in angiographic techniques. Standard techniques for placement of vascular access sheaths, angiographic catheters, and wire guides should be employed. Beacon Tip Sizing Catheters have marker bands that can be used for anatomical measurements.

SUMMARY:
This prospective observational post-market clinical study will collect data in the United States to primarily support the re-launch of the re-designed Beacon Tip Sizing Catheter and Slip-Catheter Beacon Tip Catheter & Shuttle Select Slip-Catheter (Visceral and Cerbral) for a Conformité Européenne (CE) Mark application in the European Union (EU). Additionally, the data from this study may be used to support regulatory approval in other countries/regions.

The purpose of this clinical study is to evaluate the safety and performance of these catheters in accordance with the Intended Use through the end of index procedure, and through 30 days post procedure, (as applicable as data is available) to ensure an acceptable benefit:risk ratio.

ELIGIBILITY:
Inclusion Criteria:

* A patient is deemed suitable for inclusion in this study if the patient undergoes a procedure using an applicable Beacon Tip Catheter.

Exclusion Criteria:

* Patient or his/her legally authorized representative objects to collection and processing of his/her data, or not willing to accept the use of an Informed Consent waiver or the data protection notice (if utilized).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population for this study will be patients receiving care at the 8 office-based labs (OBLs) consisting of 14 sites, all part of the Data Collection Center, Vascular Breakthroughs. These patients will not be constrained to a specific demographic, but rather will be any person who undergoes a procedure using a Beacon Tip Catheter(s).
Sampling Method: Non-Probability Sample
Enrollment: 588 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful navigation to the intended location | Duration of the procedure (approx. 1 hour)
  The primary performance outcome is successful navigation to the intended location
  The percent of successful navigation to the intended location
Successful intended use | Duration of the procedure (approx. 1 hour)
  Successful intended use (e.g. release of contrast agent (if applicable), successful anatomical sizing (if applicable)), after successful navigation to the intended location
Freedom from catheter-related major complications | up to 30 days
  The primary safety outcome is freedom from catheter-related major complications. Major complications are defined as those that:
  * Require therapy, minor hospitalization (<48 hours);
  * Require major therapy, unplanned increase in level of care, prolonged hospitalization;
  * Have permanent adverse sequelae; or result in death.
  The percent of patients with freedom from catheter-related major complications

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular Breakthroughs, Darien, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request immediately after approval or clearance of the product and ending 5 years after approval or clearance. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.